CLINICAL TRIAL: NCT04690140
Title: Can Modified Coronally Advanced Tunnel be an Alternative to Epithelialized Free Gingival Graft Technique in Gingival Phenotype Modification? A Comparative Controlled Randomized Clinical Trial
Brief Title: Can Modified Coronally Advanced Tunnel be an Alternative in Gingival Phenotype Modification?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Gencay Keceli, Assoc. Prof. Dr., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Phenotype Modification
Record Dates: First submitted 2020-12-17; First posted 2020-12-30 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2020-12

CONDITIONS: Gingival Phenotype

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients were randomly assigned into modified coronally advanced tunnel (n=25) and epithelialized free gingival graft (n=25) groups by one of the authors with an allocation ratio of 1:1 by using a computer-generated program after successful completion of phase I periodontal treatment. One calibrated author masked to the applied surgical technique recorded all clinical variables. The labeled envelope containing the intervention name was opened by the surgeon.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- modified coronally advanced tunnel technique (Active Comparator): Initial sulcular incisions and flap separation were then carried out with tunnel knives. Dissection was extended at least 8 mm apically to the mucogingival junction and the muscle attachments were removed with curettes so that the flap could be moved in a coronal direction without tension. Interdental papillae were undermined to prepare the bed for connective tissue graft placement. Connective tissue graft was then inserted under the tunnel at the sites of recession and retracted laterally by sutures towards each end of the tunnel. After connective tissue graft positioning, the flap was gently stretched coronally to obtain passive flap closure. The exposed connective tissue was covered by connecting the adjacent flap margins with additional sutures.
  Interventions: Procedure: Modified coronally advanced tunnel technique
- epithelialized free gingival graft (Active Comparator): A partial-thickness flap was elevated (blade #15c) with horizontal incisions at the cemento-enamel junction level of the adjacent teeth. Then, two vertical incisions extending to the apical were made from two ends of the horizontal incision. The epithelium in the framed region was removed with a scalpel and the underlying connective tissue was exposed. To achieve the best vascularization from the recipient site, bed preparation was completed with a split-thickness horizontal incision that joins the vertical incisions in the apical region.
  Interventions: Procedure: Epithelialized free gingival graft

INTERVENTIONS:
Procedure: Epithelialized free gingival graft — The Epithelialized free gingival graft placed on the prepared bed.
  Arms: epithelialized free gingival graft
Procedure: Modified coronally advanced tunnel technique — Connective tissue graft placed under the prepared tunnel
  Arms: modified coronally advanced tunnel technique

SUMMARY:
In the randomized comparative controlled trial, 50 patients with insufficient keratinized tissue at the anterior mandible were treated with either Modified coronally advanced tunnel or epithelialized free gingival graft. At baseline, 6th week, 6th month, 12th-month visits; keratinized tissue height, gingival thickness, recession depth, recession width, probing depth, and clinical attachment level, were evaluated. Keratinized tissue change, Gingival thickness change, root coverage, clinical attachment gain, and complete root coverage were calculated. Wound healing index, tissue appearance, patient expectations, aesthetics, and dentine hypersensitivity were assessed at baseline and 6th week.

ELIGIBILITY:
Inclusion Criteria:

* presence of at least two anterior mandibular teeth with keratinized tissue height≤1 mm with gingival thickness ≤1mm
* presence of at least two recession type-1 recessions at mandibular anterior teeth and at least one recession with recession depth ≥2 mm,
* aged between 18-60.

Exclusion Criteria:

* unstable endodontic conditions or presence of any restoration/abrasion,
* tooth mobility, any surgical history or gingival enlargement in the area,
* smoking or alcohol use,
* uncontrolled systemic disease, pregnancy or use of drugs known to affect gingival conditions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-05-05 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
Gingival Thickness | Baseline
  GT, measured at the midpoint location between the gingival margin and mucogingival junction, using an endodontic spreader (#25 endodontic spreader, 25 mm; D-perfect, Shenzhen, China).
Gingival Thickness (GT) | 6th week
  GT, measured at the mid-point location between the gingival margin and mucogingival junction, using an endodontic spreader (#25 endodontic spreader, 25 mm; D-perfect, Shenzhen, China).
Gingival Thickness (GT) | 6th month
  GT, measured at the mid-point location between the gingival margin and mucogingival junction, using an endodontic spreader (#25 endodontic spreader, 25 mm; D-perfect, Shenzhen, China).
Gingival Thickness (GT) | 12th month
  GT, measured at the mid-point location between the gingival margin and mucogingival junction, using an endodontic spreader (#25 endodontic spreader, 25 mm; D-perfect, Shenzhen, China).
Keratinized Tissue Height (KTH) | Baseline
  KTH, measured from gingival margin to the mucogingival junction (MGJ).
Keratinized Tissue Height (KTH) | 6th week
  KTH, measured from gingival margin to the mucogingival junction (MGJ).
Keratinized Tissue Height (KTH) | 6th month
  KTH, measured from gingival margin to the mucogingival junction (MGJ).
Keratinized Tissue Height (KTH) | 12th month.
  KTH, measured from gingival margin to the mucogingival junction (MGJ).

SECONDARY OUTCOMES:
Recession Depth (RD) | Baseline
  RD, measured from the cemento-enamel junction (CEJ) to the most apical extension of the gingival margin.
Recession Depth (RD) | 6th week
  RD, measured from the cemento-enamel junction (CEJ) to the most apical extension of the gingival margin.
Recession Depth (RD) | 6th month
  RD, measured from the cemento-enamel junction (CEJ) to the most apical extension of the gingival margin.
Recession Depth (RD) | 12th month.
  RD, measured from the cemento-enamel junction (CEJ) to the most apical extension of the gingival margin.
Recession width (RW) | Baseline
  Recession width (RW), the distance between the mesial gingival margin and the distal gingival margin of the tooth measured from the widest point of the recession.
Recession width (RW) | 6th week
  Recession width (RW), the distance between the mesial gingival margin and the distal gingival margin of the tooth measured from the widest point of the recession.
Recession width (RW) | 6th month
  Recession width (RW), the distance between the mesial gingival margin and the distal gingival margin of the tooth measured from the widest point of the recession.
Recession width (RW) | 12th month.
  Recession width (RW), the distance between the mesial gingival margin and the distal gingival margin of the tooth measured from the widest point of the recession.
Probing pocket depth (PD) | Baseline
  Probing pocket depth (PD), measured from the gingival margin to the bottom of the gingival sulcus.
Probing pocket depth (PD) | 6th week
  Probing pocket depth (PD), measured from the gingival margin to the bottom of the gingival sulcus.
Probing pocket depth (PD) | 6th month
  Probing pocket depth (PD), measured from the gingival margin to the bottom of the gingival sulcus.
Probing pocket depth (PD) | 12th month.
  Probing pocket depth (PD), measured from the gingival margin to the bottom of the gingival sulcus.
Clinical attachment level (CAL) | Baseline
  Clinical attachment level (CAL), measured from the cementoenamel junction to the bottom of the gingival sulcus.
Clinical attachment level (CAL) | 6th week
  Clinical attachment level (CAL), measured from the cementoenamel junction to the bottom of the gingival sulcus.
Clinical attachment level (CAL) | 6th month
  Clinical attachment level (CAL), measured from the cementoenamel junction to the bottom of the gingival sulcus.
Clinical attachment level (CAL) | 12th month
  Clinical attachment level (CAL), measured from the cementoenamel junction to the bottom of the gingival sulcus.
Keratinized tissue change (KTC) | Baseline
  Keratinized tissue change (KTC), GT change (GTC), root coverage, clinical attachment gain (CAG) were calculated in millimeters and percentages.
Keratinized tissue change (KTC) | 6th week
  Keratinized tissue change (KTC), GT change (GTC), root coverage, clinical attachment gain (CAG) were calculated in millimeters and percentages.
Keratinized tissue change (KTC) | 6th month
  Keratinized tissue change (KTC), GT change (GTC), root coverage, clinical attachment gain (CAG) were calculated in millimeters and percentages.
Keratinized tissue change (KTC) | 12th month
  Keratinized tissue change (KTC), GT change (GTC), root coverage, clinical attachment gain (CAG) were calculated in millimeters and percentages.
Wound healing index (WHI) | 6th week
  Wound healing index (WHI) was recorded two-weeks after surgery. The wound surface was visually inspected and the soft tissue healing was defined as 'uneventful' (score 1), 'slightly disturbed' (score 2) or 'poor' (score 3) based on the presence and severity of the items including patient discomfort, erythema, edema, suppuration and flap dehiscence.
Tissue appearance (TA) | 6th week
  Tissue appearance (TA) was evaluated by asking the patients to score the consistency, contour, color match, keloid formation degree and contiguity of their treated sites at T2. The scores were collected as points, shown in parentheses, by asking the consistency as firm (1p) or spongy (0p); contour as presence (2p) or absence (0p) of knife-edged and scalloped gingival margin; color match as excellent (3p), good (2p), adequate (1p) or unsatisfactory (0p); keloid formation degree as absent (1p) or present (0p); contiguity as the presence (-1p) or absence (0p) of each perceptible incision mark.
Dentine hypersensitivity (DH) | 6th week
  Dentine hypersensitivity (DH) was evaluated with air evaporative stimulus method at baseline and T2. After placement of finger(s) for preserving the nearby teeth, the recession sites were subjected to evaporative stimulus comprised of 1-second air blast from 1 to 3 mm distance by using the air spray at 40-65 psi pressure and 19±50C. After application, the patients were requested to give a score to their DH between 0 (=no pain) and 10 (=extreme pain).
Patient expectations (PE) | 6th week
  Patient expectations (PE) were evaluated by requesting from the patients to rate their treatment results at T2, as satisfactory or not, in terms of appearance, experience and obtained root coverage.
Aesthetics (A) | 6th week
  Aesthetics (A) was evaluated by the patient at T1 by rating its level as excellent, good, fair or poor.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Yilmaz BT, Comerdov E, Kutuk C, Nart J, Keceli HG. Modified coronally advanced tunnel versus epithelialized free gingival graft technique in gingival phenotype modification: a comparative randomized controlled clinical trial. Clin Oral Investig. 2022 Oct;26(10):6283-6293. doi: 10.1007/s00784-022-04580-0. Epub 2022 Jun 16. PMID 35708779